CLINICAL TRIAL: NCT01059656
Title: A Phase IIa Open Multicenter, Trial, of Treatment With Pazopanib (Multi Tyrosine Kinase Inhibitor) in Dermatofibrosarcomas (DFSP), Unresectable Locally Advanced (Potentially Mutilating Surgery), Primary or Relapsing , Transformed or Not.
Brief Title: Phase II Pazopanib Study in Advanced Dermatofibrosarcomas
Acronym: DFSP-PAZO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision of Study Principal Investigator
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P090402; 2009-014096-46 (EudraCT Number)
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Dermatofibrosarcomas of DARIER FERRAND(DFSP)
Keywords: Dermatofibrosarcoma; Pazopanib¨; Phase II
MeSH Terms: conditions — Dermatofibrosarcoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1:Pazopanib (Experimental): Pazopanib 800mg/j
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Administration of pazopanib per os 800mg/ qd during 6 months until stable response according to primary endpoint, with 3 monthly successive examinations, and for a period of study not exceeding 18 months.

SUMMARY:
In relation to the activation of PDGF-mediated signalization due to the fusion gene COL1A1-PDGFb in DFSP, imatinib (800mg/day) has shown activity in advanced DFSP and has became the reference treatment option for these patients. Yet the activity observed does not allow for a downstaging compatible with successful resection in a number of patients and does not prevent subsequent tumour progression in case of residual tumour.Pazopanib in relation to 1) its multi tyrosine kinase inhibiting activity (VEGFR-1, VEGFR-2, VEGFR-3, PDGFR-α, PDGFR-β and c-kit with IC50 values of 10, 30, 47, 71, 84, and 74 nM, respectively) involving in particular PDGFR, and VEGFR which has been shown to be activated in DFSP, 2) its antitumour activity in sarcomas patients, and 3) its acceptable safety profile, is a logical candidate for therapeutic trials in DFSP both in patients not expected to derive a sufficient benefit from imatinib and in patients failing imatinib mesylate. Moreover, using quantitative RT-PCR and immunohistochemistry we have recently demonstrated high levels of VEGF and VEGFR2 expression in dermatofibrosarcoma.

DETAILED DESCRIPTION:
Dermatofibrosarcoma protuberance (DFSP) is a rare soft tissue sarcoma of intermediate malignant potential. Treatment relies on a wide local excision with negative margin and with frequent need of reconstructive surgery. A translocation between chromosomes 17 and 22 that places the platelet-derived growth factor-B (PDGFB) under the control of the collagen 1A1 promoter is present in > 90 % of the cases leading to an up regulation of PDGF-β expression and activation of the tyrosinase kinase PDGFRβ. Imatinib mesylate has been approved in unresectable and metastatic DFSP due to its activity on PDGFR. This study will evaluate the benefit of pazopanib, a multikinase inhibitor in advanced DFSP. Administration of pazopanib per os 800mg/ qd during 6 months until stable response according to primary endpoint , and for a period of study not exceeding one year.In case of progression evaluated according to the primary endpoint after a period of treatment superior to one month, or in the absence of response at 3 months, the patient will be withdrawn from study, in order to get alternative therapeutics. These patients will be considered as failures for analysis. After a 6-month treatment period, and reaching a stable response, treatment continuation decision will be based on the operability of patients.

Administration of pazopanib per os 800mg/ qd during 6 months until stable response according to primary endpoint, with 3 monthly successive examinations, and for a period of study not exceeding 18 months.In case of progression evaluated according to the primary endpoint after a period of treatment superior to one month, or in the absence of response at 3 months, the patient will be withdrawn from study, in order to get alternative therapeutics. These patients will be considered as failures for analysis. After a 6-month treatment period, and reaching a stable response, treatment continuation decision will be based on the operability of patients Statistical analysis : The trial has been planned using a one-stage design (Fleming TR. Et al) Analysis of the main endpoint will rely on a one-sided binomial test comparing the observed response rate to the expected response rate under the null hypothesis . The type I error rate is fixed at 0.025.For the main endpoint, a point estimate and a two-sided 90% confidence interval will be presented, which will be consistent with the one-sided test at a 0.025 level. For secondary endpoints, point estimates and 95% confidence intervals will be presented.We intend to estimate the probability of tumour size reduction of at least 30%. The sample size was calculated by FLEMMING method : Ho will be defined by a RR ≤20% (decrease in tumour size of at least 30%) , H1 , response rate, 26 patients must be included in order to demonstrate an efficacy as defined by a RR≥50%, with a 90% power and alfa 2.5% one side.

ELIGIBILITY:
Inclusion Criteria:

* Primitive unresectable DFSP, locally advanced (potentially mutilating surgery), or in relapse or transformed.
* Histologic confirmation of the Darier-FERRAND tumour (transformed types will be accepted provided a previous caryotype confirming the translocation (17,22)
* Age > or equal to 20 years
* Signed informed consent
* Appropriate contraception
* No evolutive tumoural disease except baso-cellular carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.

Exclusion Criteria:

* Patient refusal to participate
* Age < 20 years
* Pregnant or lactating women
* Other evolutive tumour disease except baso-cellular carcinoma
* Haematologic abnormalities:Hemoglobin < 9g/dl, PNN <
* 1500/mm3, Platelets <100000/mm3
* AST and ALT > 2N
* Bilirubin > 1.5N
* Creatinin > 1.5mg/dL or creatinin clearance <30ml/mn
* Proteinuria >1g/24h
* Serum albumin< 2.5g/dL
* Hepatitis B, C and/or HIV known Infection
* Treatment interfering with pazopanib
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks prior to beginning therapy, or anticipation of the need for a major surgical procedure during the course of the study.
* Clinically significant gastrointestinal abnormalities including, but not limited to:Malabsorption syndromeDisease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect the absorption of study drug.Active peptic ulcer diseaseInflammatory bowel diseaseUlcerative colitis, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis or other gastrointestinal condition increasing the risk of perforation.History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment· Presence of active or uncontrolled infection.
* Evidence of active bleeding or bleeding diathesis.
* History of any one or more of the following cardiovascular conditions within the past 6 months:Coronary/peripheral artery bypass graft, cardiac angioplasty or stenting.Myocardial infarction.Severe/unstable angina pectoris.Symptomatic peripheral vascular disease pulmonary embolism, thromboembolic event, cerebrovascular accident or transient ischemic attack.Class III or IV congestive heart failure, as defined by the New York Heart Association
* Cardiovascular disease with NYHA > II
* Poorly controlled hypertension (defined as a systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) ≥90 mmHg.
* Following abnormalities on ECG : Q wave, ischemia, QTc > 450 msec, atrioventricular block 2 or 3, atrial fibrillation
* Therapeutic anticoagulation treatment.
* Chronic daily treatment with aspirin (≥ 100 mg/day) or non-steroidal anti-inflammatory agents known to inhibit platelet function. Treatment with dipyridamole, ticlopidine, clopidogrel and/or cilostazol is also not allowed.. Concurrent treatment with an investigational agent or participation in another clinical trial.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib.
* Taken by the order treatment anti cancerous concomitants within 4 weeks previous inclusion
* Radiotherapy on the hurt within 3 months previous inclusion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Decrease of at least 30% of the biggest diameter measured clinically at 6 months preceded by clinical response | at 3 months

SECONDARY OUTCOMES:
For measure of tumour volume : Measure of radiologic response (" MULTIBARETTE " MDCT scanner) using RECIST criteria and OMS (WHO) | at 3 months
For measure of tumour volume : Measure of the volume of the tumour (" MULTIBARETTE " MDCT scanner) in each centre | at 3 months
For measure of tumour volume : Research of translocation COL1A1-PDGFB by FISH (paraffin) and caryotype on fresh tissue (centralisation in F PEDEUTOUR laboratory, Nice) | at 3 months
Prognostic factors of tumoral response : Semi-quantitative measure of apoptosis on surgical piece and of senescence | at inclusion, M1, M3 and M6
Expression of the phosphorylated form of the receptors of PDGFB and VEGF and of the MAPK. | at inclusion, M1, M3 and M6
Prognostic factors of tumoral response :Clinical and biologic safety Common Terminology Criteria forAdverse Events v3.0 (CTCAE) | at every visit except M0
Prognostic factors of tumoral response :Evaluation of QOL, EORTC QLQ-C30 | M0, M3, M6, M9, M12, M15 and M18

CONTACTS AND LOCATIONS:
Overall Officials: Celeste LEBBE, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint-Louis - Service de Dermatologie (Pole POPS), Paris, France

REFERENCES:
- [Derived] Delyon J, Porcher R, Battistella M, Meyer N, Adamski H, Bertucci F, Guillot B, Jouary T, Leccia MT, Dalac S, Mortier L, Ghrieb Z, Da Meda L, Vicaut E, Pedeutour F, Mourah S, Lebbe C. A Multicenter Phase II Study of Pazopanib in Patients with Unresectable Dermatofibrosarcoma Protuberans. J Invest Dermatol. 2021 Apr;141(4):761-769.e2. doi: 10.1016/j.jid.2020.06.039. Epub 2020 Sep 18. PMID 32956651